CLINICAL TRIAL: NCT01143220
Title: Japanese Assessment of Indication Based Programming
Acronym: JASMINE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Guidant Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: JASMINE 0709
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure; Arrhythmias, Cardiac
Keywords: Cardiac Resynchronization Therapy; Heart Failure; Pathologic Processes; Heart Diseases; Tachycardia; Cardiovascular Diseases; Ventricular Flutter; Tachycardia, Ventricular; Ventricular Fibrillation; Arrhythmias, Cardiac; Ease of Use
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac; Pathologic Processes; Heart Diseases; Tachycardia; Cardiovascular Diseases; Ventricular Flutter; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD / CRT-D patient: Patients implanted with a single or dual chamber ICD or CRT-D device approved in Japan capable of using the IBP feature.
  Interventions: Other: No specific interventions

INTERVENTIONS:
Other: No specific interventions — Observational investigation, only procedures according to local hospital standard.

SUMMARY:
The purpose of this clinical investigation is to assess the programming behavior of the physicians in the patient cohort. Furthermore, the acceptance level of specific programming recommendations based on the patient's clinical needs and primary indications will be evaluated by comparing parameters determined by the feature IBP to daily life programming chosen by physicians.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a single or dual chamber ICD or CRT-D device approved in Japan capable of using the IBP feature.
* Geographically stable patients who are available for follow-up at a study center .
* Age 20 years or above.
* Patients, who do receive all leads that are supposed to be used with a certain type of device (i.e. no dual chamber ICD / CRT-D device without an atrial lead or CRT-D devices with only one ventricular lead).

Exclusion Criteria:

* Inability or refusal of the patient to give approval to collect/store/process personal health information at the sponsor.
* Pregnant women or women, planning to become pregnant .
* Any kind of previous CRM device therapy (no replacements, no upgrades, no new implants after complete system removals ).
* Enrolment in another clinical trial or clinical investigation without prior notification of the sponsor .
* Estimated life expectancy of less than six months per judgment of the physician.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population comprises the standard patient population of the participating sites indicated for the intended devices per local guidelines in the study centers.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that are programmed by the physician to anything other than the specific IBP parameter settings | Enrollment / Last available follow up during the first six months after implant
  The primary endpoint is the proportion of patients that are programmed by the physician to anything other than the specific IBP parameter settings determined for the particular patient. The specific IBP parameter set is determined either by the physician using the IBP feature or by creating the most appropriate set of IBP parameters using the information given in the patient history section of the CRF. Each IBP recommended parameter will be evaluated individually.

SECONDARY OUTCOMES:
Degree of acceptance of IBP | Enrollment / Last available follow up during the first six months after implant
  Measured by a composite endpoint on a 0 to 100 scale, reflecting all parameter changes for each patient between the IBP recommended parameter set and finally programmed parameter set of the last recorded visit. The impact on the endpoint will vary by the parameter reprogrammed. Weights will be determined for each parameter based upon the relevance of the parameter to the overall acceptance of the IBP algorithm.
Proportion of patients without any IBP use | First six months after implant.
Proportion of patients without any IBP use at enrollment, but IBP use during follow up. | First six months after implant.
Proportion of patients with IBP use only at enrollment. | First six months after implant.
oProportion of patients with IBP use during enrollment and additional subsequent use of IBP during follow up. | First six months after implant.
Proportion of parameters changed per patient from nominal device settings. | First six months after implant.
Proportion of parameters changed per patient from IBP recommended device settings, if IBP was used. | First six months after implant.
Differences between nominal parameters and final programming by physicians for parameters with quantitative values. | First six months after implant.
Differences between parameters recommended by IBP and final programming by physicians for parameters with quantitative values | First six months after implant.
Total number of parameter changes recorded during the enrollment procedure after IBP recommendations were programmed. | First six months after implant.
Total number of parameter changes to a value different from the device nominals recorded during the enrollment procedure | First six months after implant.
oTotal number of parameter changes during follow up procedure(s) | First six months after implant.
Frequency of changes made to a single parameter during the time the patient is enrolled in the clinical investigation. | First six months after implant.

CONTACTS AND LOCATIONS:
Locations (45):
- Japan (45):
  - Social Insurance Chukyo Hospital, Nagoya, Aichi-ken
  - Hiraka General Hospital, Yokote, Akita
  - Kameda Medical Hospital, Kamogawa, Chiba
  - Shin-Tokyo Hospital, Matsudo, Chiba
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Saiseikai Imabari Hospital, Imabari, Ehime
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Aso Iizuka Hospital, Iizuka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Shinkoga Hospital, Kurume, Fukuoka
  - Shinsapporo Hospital of Cardiology, Sapporo, Hokkaido
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Hokkaido Social Insurance Hospital, Sapporo, Hokkaido
  - Hokkaido Medical Center, Sapporo, Hokkaido
  - Hokko Memorial Hospital, Sapporo, Hokkaido
  - Kanazawa Cardiovascular Hospital, Kanazawa, Ishikawa-ken
  - Tokai University Hospital, Isehara, Kanagawa
  - Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Kumamoto Central Hospital, Kumamoto, Kumamoto
  - Kyoto Katsura Hospital, Kyoto, Kyoto
  - Kyoto Prefectual University of Medicine Hospital, Kyoto, Kyoto
  - Uji Tokushukai Hospital, Uji, Kyoto
  - Yamada Red Cross Hospital, Ise, Mie-ken
  - Matsumoto Kyoritsu Hospital, Matsumoto, Nagano
  - Nagano Chuo Hospital, Nagano, Nagano
  - Nagano Red Cross Hospital, Nagano, Nagano
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Iseikai Hospital, Osaka, Osaka
  - Kinki University Hospital, Sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Hamamatsu Medical Center, Hamamatsu, Shizuoka
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Shizuoka Hospital, Izunokuni, Shizuoka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - Juntendo University Hospital, Tokyo, Tokyo
  - The University of Tokyo Hospital, Tokyo, Tokyo
  - Tokyo Women's Medical University Medical Center East, Tokyo, Tokyo
  - Tokyo Heart Center Osaki Hospital, Tokyo, Tokyo
  - Toho University Ohashi Medical Center, Tokyo, Tokyo
  - Keio University Hospital, Tokyo, Tokyo
  - Ogikubo Hospital, Tokyo, Tokyo
  - Yamaguchi Grand Medical Center, Hōfu, Yamaguchi
  - Yamaguchi-ken Saiseikai Shimonoseki General Hospital, Shimonoseki, Yamaguchi